CLINICAL TRIAL: NCT05812989
Title: Modifiers and Mechanisms of Loneliness Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathi Heffner, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007800; P30AG064103-Pilot7 (Other Grant/Funding Number: Rochester Roybal Center for Social Ties & Aging Research); P30AG064103 (NIH)
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Loneliness
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Engage Coaching (Active Comparator): Social Engage Coaching involves psychoeducation on the importance of social connections for health as well as structured goal setting and problem solving for increasing social connectedness.
  Interventions: Behavioral: Social Engage Coaching
- Social Engage Coaching with Connect for Caregivers (Active Comparator): Social Engage Coaching involves psychoeducation on the importance of social connections for health as well as structured goal setting and problem solving, guided by use of a digitized prioritization tool, for increasing social connectedness.
  Interventions: Behavioral: Social Engage Coaching; Behavioral: Connect for Caregivers

INTERVENTIONS:
Behavioral: Social Engage Coaching — Participants will complete up to 8 weekly individual Social Engage psychotherapy sessions. Participants will be allotted up to 3 months to complete all sessions, a time-frame that allows for two weeks without meeting to address life stressors such as illnesses that may pop up. All sessions are provided via phone or videocall (Zoom). The first and last session are longer - up to 60 minutes if needed. Middle sessions are shorter (20-45 minutes). Engage is a stepped care psychotherapy in that the simplest strategy is taught first-action planning (a derivative of problem solving therapy)-and "barrier strategies" are added only if needed. Action plans are designed to address loneliness and social isolation in the context of caregiving demands.
Behavioral: Connect for Caregivers — Participants will complete an individual session with a coach who will use a digitized prioritization tool to help identify goals and an action plan for social connectedness.
  Other Names: Digitized prioritization of goals and action planning for social engagement.
  Arms: Social Engage Coaching with Connect for Caregivers

SUMMARY:
A specific aim of this research is to identify the role of emotion regulation in response to social threat in caregivers' response to a behavioral coaching intervention for loneliness. A second aim of the study is to determine the benefit of a digitized, social engagement prioritization tool for improving coaches' intervention fidelity and caregiver outcomes. This study is funded through the Pilot Award Program of the Rochester Roybal Center for Social Ties & Aging Research, a UR Center funded by the National Institute on Aging by grant P30AG064103.

DETAILED DESCRIPTION:
The objective of this Stage III mechanistic study is to help identify additional modifiable targets and scalable approaches to support further development of highly effective, mechanistic-informed approaches to reducing loneliness and improving social connectedness in caregivers. This study is a Stage III, 19-month 2 (groups) x 2 (assessment timepoints) randomized clinical trial (RCT) aimed at identifying whether lonely caregivers' capacity, is associated with the degree to which loneliness is reduced in response to social engagement intervention (S-ENG). Further, the study will address whether a digitized, social engagement prioritization tool (C4C) used in the first session of S-ENG can improve intervention fidelity and

ELIGIBILITY:
Inclusion Criteria:

* Caregiver (age 50 or older) for a community-dwelling loved one with Alzheimer's disease or related dementia (ADRD), living with (or in close proximity to) the person with ADRD.
* Elevated caregiving distress: above population mean (>11) on 10-item Perceived Stress Scale (PSS-10) and/or at least moderate caregiver strain (score >= 5) on the Modified Caregiver Strain Index.
* Social disconnection: UCLA Loneliness Scale: Short Form score of > 5.

Exclusion Criteria:

* Non-English speaking
* Significant cognitive impairment
* Major cardiovascular conditions that may interfere with reliable assessment of HRV (e.g., congestive heart failure, pacemaker, prior myocardial infarction).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Loneliness | 11 weeks
  UCLA Loneliness Scale Version 3, which assesses self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. However, some individual items must be reverse-coded so that higher total scores reflect greater loneliness (i.e., 1=4, 2=3, 3=2, 4=1). These items (e.g., "How often do you feel there are people you can turn to?") are items 1,5,6,9,10,15,16,19,20. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness).
High frequency heart rate variability (HF-HRV) | 11 weeks
  HF-HRV is derived by spectral analysis of the electrocardiograph (ECG) waveform collected during a rest period, and is a measure of parasympathetic control of the heart; Higher resting HF-HRV (absolute power of the high-frequency band (0.15-0.4 Hz) in ms-squared) reflects greater parasympathetic regulation of the heart.
Dot probe task | 11 weeks
  Difference in response times (in milliseconds) to dots appearing in the location of a previously shown negative versus the neutral face.
Affect (valence) from Self-Assessment Manikin | 11 weeks
  Mean valence score during negatively valenced social pictures. The Self-Assessment Manikin is a non-verbal pictorial assessment technique that directly measures a person's affect in response to positive, negative, and neutrally valenced pictures. Affect valence is measured on a 9-point scale: 1 (very unpleasant) - 9 (very pleasant).
Stroop Task | 11 weeks
  Difference in response time (ms) to judgments of semantic meaning (positive or negative) of spoken, socially-relevant words between congruent (e.g., negative social word-negative vocal tone) versus incongruent (e.g., positive social word-negative vocal tone) trials, indicating cognitive interference.

SECONDARY OUTCOMES:
Flanker Task | 11 weeks
  During the trials, a decision needs to be made about whether the orientation of a central stimulus is congruent or incongruent with a set of flanking arrows. Selective attention/cognitive inhibition is indicated by difference between response time (millisecond) on the congruent and incongruent conditions.
Set-Shifting Task | 11 weeks
  During each trial, the participant is required to match a stimulus on the top of the screen to one of two stimuli in the lower corners of the screen. In task-homogeneous blocks, the examinee performs either Task A (e.g., classifying shapes) or Task B (e.g., classifying colors). In task-heterogeneous blocks, the examinee alternates between the two tasks pseudo-randomly. Cognitive flexibility (or capacity for task switching) is derived as the difference in response time (milleseconds) between homogeneous and heterogenous blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Kathi L Heffner, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and health history data from assessments with 57 older adults who are caregivers for individuals with ADRD. Data from this research will be made available to the public in the University of Rochester's institutional repository, UR Research, at https://urresearch.rochester.edu. We will share the research protocols, in a text format, such as MS Word or PDF. Any qualitative data will also be made available in text form. For quantitative data, the PI will make available the actual datasets generated from research, in a commonly- used format such as a SAS® dataset. The datasets will be associated with a related publication, research protocol or other documentation of the original research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Timetable to release the data: the data and referenced resources from publications will be made available by the on-line publication date.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement as suggested by the NIH that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. 4. De-identification of data from human subjects: A final complete database will be created to host all data which will be stripped of any identifiers and stored pursuant to UR Institutional Review Board protocols. Confidentiality for research subjects for qualitative data will be promoted by the use of an anonymization scheme and anonymizing the data as the qualitative files are created for the analysis (following guidelines developed by the Inter-university Consortium for Political and Social Research, 2012).
URL: https://urresearch.rochester.edu